CLINICAL TRIAL: NCT00874588
Title: Phase I Trial in Studying Peptide Vaccine Therapy Targeting to Cancer Specific Antigen Combined With Anti-angiogenic Peptide Antigen in Treating Patients With Advanced or Recurrent Non-small Cell Lung Cancer
Brief Title: Peptide Vaccine Targeting to Cancer Specific Antigen Combined With Anti-angiogenic Peptide Antigen in Treating Patients With Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fukushima Medical University (Other)
Collaborators: Human Genome Center, Institute of Medical Science, University of Tokyo (Other)
Responsible Party: Principal Investigator, Hiroyuki Suzuki, Professor, Fukushima Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FVT-L0901
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — NUF2 protein, human; Receptor Protein-Tyrosine Kinases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phase I study (Experimental)
  Interventions: Biological: HLA-A*2402restricted URLC10, CDCA1, VEGFR1 and VEGFR2

INTERVENTIONS:
Biological: HLA-A*2402restricted URLC10, CDCA1, VEGFR1 and VEGFR2 — Escalating doses of every peptide will be administered by subcutaneous injection on days 1,8,15 and 22 of each 28-day treatment cycles. Planned doses of peptides are 1.0mg and 3.0mg.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, immune response and clinical response of different doses of HLA-A*2402 restricted epitope peptides URLC10, CDCA1, VEGFR1 and VEGFR2 emulsified with Montanide ISA 51.

DETAILED DESCRIPTION:
URLC10 and CDCA1 have been identified as cancer specific molecules especially in non small cell lung cancer using genome-wide expression profile analysis by cDNA microarray technique. We have determined the HLA-A*2402 restricted epitope peptides derived from these molecules. We also tend to use the peptides targeting to tumor angiogenesis. VEGF receptor 1 and 2 are essential targets to tumor angiogenesis, and we identified that peptides derived from these receptors significantly induce the effective tumor specific CTL response in vitro and vivo. According to these findings, in this trial, we evaluate the safety, immunological and clinical response of those peptides.

ELIGIBILITY:
Inclusion Criteria:

Disease characteristics

1. Advanced or recurrent non small cell lung cancer
2. Second line or later therapeutic status

Patient characteristics

1. ECOG performance status 0-2
2. Life expectancy > 3 months
3. HLA-A*2402
4. Laboratory values as follows 1500/mm3<WBC<15000/mm3 Platelet count>75000/mm3 Bilirubin < 3.0mg/dl Asparate transaminase < 99IU/L Alanine transaminase < 126IU/L Creatinine < 2.2mg/dl
5. Able and willing to give valid written informed consent

Exclusion Criteria:

1. Active and uncontrolled cardiac disease (includes patients with myocardial infarction within 6 months before entry)
2. Pregnancy (woman of child bearing potential)
3. Active and uncontrolled infectious disease
4. Adrenal cortical steroid hormone dependent status
5. Decision of unsuitableness by principal investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Adverse effects, dose limiting toxicity, and maximum tolerated dose as measured by CTCAE ver3.0 pre treatment, during study treatment, and 3 months after treatment | 3 months

SECONDARY OUTCOMES:
Peptides specific CTL responses in vitro | 3 months
Objective response rate as assessed using RECIST criteria | 6 months
Changes in levels of regulatory T cells | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fukushima Medical University, Fukushima, Japan

REFERENCES:
- [Background] Ishizaki H, Tsunoda T, Wada S, Yamauchi M, Shibuya M, Tahara H. Inhibition of tumor growth with antiangiogenic cancer vaccine using epitope peptides derived from human vascular endothelial growth factor receptor 1. Clin Cancer Res. 2006 Oct 1;12(19):5841-9. doi: 10.1158/1078-0432.CCR-06-0750. PMID 17020992
- [Background] Wada S, Tsunoda T, Baba T, Primus FJ, Kuwano H, Shibuya M, Tahara H. Rationale for antiangiogenic cancer therapy with vaccination using epitope peptides derived from human vascular endothelial growth factor receptor 2. Cancer Res. 2005 Jun 1;65(11):4939-46. doi: 10.1158/0008-5472.CAN-04-3759. PMID 15930316
- [Background] Hayama S, Daigo Y, Kato T, Ishikawa N, Yamabuki T, Miyamoto M, Ito T, Tsuchiya E, Kondo S, Nakamura Y. Activation of CDCA1-KNTC2, members of centromere protein complex, involved in pulmonary carcinogenesis. Cancer Res. 2006 Nov 1;66(21):10339-48. doi: 10.1158/0008-5472.CAN-06-2137. PMID 17079454
- [Derived] Suzuki H, Fukuhara M, Yamaura T, Mutoh S, Okabe N, Yaginuma H, Hasegawa T, Yonechi A, Osugi J, Hoshino M, Kimura T, Higuchi M, Shio Y, Ise K, Takeda K, Gotoh M. Multiple therapeutic peptide vaccines consisting of combined novel cancer testis antigens and anti-angiogenic peptides for patients with non-small cell lung cancer. J Transl Med. 2013 Apr 11;11:97. doi: 10.1186/1479-5876-11-97. PMID 23578144